CLINICAL TRIAL: NCT04124783
Title: Pilot Study to Evaluate the Effects of the Nanoheath, Inc. Cooling Bolero in Women With Common Menopause Symptoms
Brief Title: Study to Evaluate the Effects of the Cooling Bolero in Women With Menopause Symptoms
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The company no longer provided the device.
Sponsor: Englewood Hospital and Medical Center (Other)
Collaborators: Nanohealth, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-19-779
Record Dates: First submitted 2019-10-10; First posted 2019-10-11 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Menopause Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cooling Bolero (Experimental)
  Interventions: Device: Cooling Bolero

INTERVENTIONS:
Device: Cooling Bolero — A vest filled with a new material (not ice or a gel) that provides controlled cooling by absorbing heat

SUMMARY:
The Cooling Bolero is a vest filled with a new material (not ice or a gel) that provides controlled cooling by absorbed heat. The vest is manufactured by Nanohealth. It intended to provide moderate cooling (~15C/59F) through indirect contact with the skin. The material in the device is safe, non-toxic, and eco-friendly.

Recent anecdotal studies of women with common peri-menopausal and menopausal symptoms (hot flashes, night sweats, flushing/sweating of face and neck, and intermittent sleep disturbances) have shown a reduction in both the frequency and intensity of those symptoms after using the Cooling Bolero. Specific (moderate) temperature cooling of the neck and upper torso appears to target and mitigate these common menopausal symptoms. This pilot study attempts to collect additional data on the effects of the Cooling Bolero.

DETAILED DESCRIPTION:
Participants who have consented for this study will first be asked to complete a Baseline Assessment of their menopausal symptoms, including documentation of their baseline weight. If the assessment indicates that the participant has at least 'moderate' menopausal symptoms, then she will then enter the Run-In Period.

During the two-week Run-In Period, participants will use a Symptom Diary for to document the frequency and severity of their menopausal symptoms. At the start of Week 3, participants will return their completed Run-In Period Symptom Diary and receive their Cooling Bolero with instructions on how to use the product during the Treatment Period.

During the Treatment Period, participants should use the Cooling Bolero at least two times per day (morning and evening) for one hour. As feasible, the participant should start to wear the product 30 minutes prior to meal time for these two applications. The participant may also wear the product at additional times, as desired. All applications of the Cooling Bolero during the four-week Treatment Period are to be documented in the Product/Symptom Diary. During the Treatment Period, the participant will also continue to document the frequency and severity of their menopausal symptoms in the Product/Symptom Diary.

At the end of Week 6, the participant will stop using the Cooling Bolero. She will be asked to complete a Product Assessment and have her weight documented.

Participants will be contacted at Week 10 to ask about the status of menopausal symptoms after four weeks of not using the Cooling Bolero

ELIGIBILITY:
Inclusion Criteria:

* Female who is at least 18 years old
* Self-reports having at least two (2) daily hot flashes associated with menopause

Exclusion Criteria:

* Taking hormonal therapy (currently or within the last 3 months).
* Has another existing medical condition that would prevent study compliance.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2020-12-23 (Actual)

PRIMARY OUTCOMES:
Number of participants with a reduction in the frequency and/or intensity of menopause symptoms | one month
  Diaries will be used to capture data pre-intervention, during the intervention, and post-intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Englewood Health, Englewood, New Jersey, United States